CLINICAL TRIAL: NCT03903978
Title: Efficacy and Effectiveness of a Self-applied Online Program to Promote Resilience and Coping Skills in University Students in Three Spanish-speaking Countries: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy and Effectiveness of a Self-applied Online Program to Promote Resilience and Coping Skills in College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Labpsitec_CORE
Record Dates: First submitted 2018-09-18; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: CORE Condition; Healthy Lifestyle Psychoeducational Program; Waiting List Control
Keywords: Resilience; University students; Prevention; Online intervention
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CORE condition (Experimental): CORE is a 6-week web-based prevention programme whose main objective is to teach coping skills and strategies to cope with stressful everyday situations in order to improve resilience, promote self-efficacy and increase well-being. The intervention consists of 6 interactive modules designed for weekly sessions and organized in 6 dimensions: autonomy, self-acceptance, environmental mastery, purpose in life, positive relationships, and personal growth. Each module includes exercises to practice the proposed skills. The program includes multimedia elements: videos, audios, vignettes, images.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Healthy lifestyle (Active Comparator): This program will provide information to promote a healthy lifestyle, on issues related to physical and mental health and physical activity, as well as diet and sleep management. The components of psychoeducation are based on the intervention protocol for depression (Castro, et al. 2015) based on low intensity psychological intervention models for mild or moderate depressive symptoms in primary care (Garcia-Herrera et al 2011; NICE, 2009; Nieuwsma et al 2012).
  Interventions: Behavioral: Healthy lifestyle
- Waiting List Control (No Intervention): Participants assigned to the Waiting List control group will be evaluated and monitored at the start of the study, 4 weeks, 8 weeks and follow-ups at 3 months. After the last follow-up evaluation, they will be given access to CORE training.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The training protocol consists of 6 weekly modules:
  0.Welcome:Introduction module to the program, with an explanation about the tools and the way to use CORE
  1. Psychoeducation: Explanation of psychological wellbeing and the concept of resilience
  2. Autonomy, building my way: Enhancement of autonomy
  3. Mindfulness and self-compassion:Training in mindfulness, savoring, and an attitude of self-compassion
  4. Overcoming obstacles: Development of coping strategies to deal with daily difficulties in life
  5. Connecting to others:Acknowledge the relevance of relationships and how they can be helpful in the construction of well-being
  6. Purpose in life and personal growth:Approach the future with a positive attitude, planning goals for the future.
  Arms: CORE condition
Behavioral: Healthy lifestyle — 1. Beginning of a lifestyle change The patient will learn to identify healthy and risky behaviors and recognize obstacles that prevent them from adopting a healthy lifestyle.
  2. Physical activity The importance of "moving on" and activating behavior will be taught through regular exercise information to improve mood.
  3. Diet This module is dedicated to teaching the importance of diet for good physical and mental health. The Mediterranean diet will be taken as an example for a balanced and balanced diet, because it does not differ from the habits of other countries.
  4. Sleep The importance of good sleep will be addressed with information and strategies for understanding the relationship between sleep and overall health.
  Arms: Healthy lifestyle

SUMMARY:
This study aims to evaluate the effectiveness and efficiency of this intervention protocol applied to three populations of Spanish-speaking university students (Spain, Argentina and Mexico). The purpose of this paper is to present the protocol designed to carry out the randomised controlled study (RCT).

DETAILED DESCRIPTION:
This study is a multi-country randomized controlled trial (RCT) with three groups comparing efficacy of unguided Internet-based intervention for students low on resilience with three conditions: a) unguided web-based resilience intervention (CORE); 2) Healthy lifestyle psychoeducationalprogram (HLP); and 3) Care as usual condition (CAU). Online- and telephone assessments will be conducted at pre- and post-intervention, and at 6- and 12-month follow-up (see Figure 1). Participants will be randomized in a 1:1 ratio. Randomization will be stratified according to trial site.

The aim of this trial is to evaluate the efficiency and effectiveness of an Internet-based programme developed to promote resilience and coping skills among at-risk university students in Spain, Argentina and Mexico. The specific aims are:

1. To provide a preventative online intervention for enhancing resilience for decreasing symptoms of depression and anxiety and for increasing wellbeing
2. To evaluate the effectiveness and acceptability of CORE program in a randomized controlled trial compared with two conditions, Healthy lifestyle (HTP) and care as usual (CAU).
3. To analyze feasible strategies to implement CORE and to identify possible implementation barriers from final users, professionals of University counseling services and the University authorities in three Spanish-speaking countries.

ELIGIBILITY:
Inclusion Criteria:

* University students with a standard deviation score below the sample mean on the Connor-Davidson Resilience Scale (CDRISC-25).
* Adequate knowledge to understand and read Spanish and/or be Spanish-speaking.
* Internet access and computer skills.

Exclusion Criteria:

* University students who are on a waiting list for psychotherapy or who are or have been undergoing psychotherapy in the last 12 months.
* Individuals with a current or past psychotic or bipolar disorder.
* Individuals at risk of suicide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Connor-Davidson's Resilience Scale (CDRISC; Connor and Davidson, 2003) | Up to 3 months
  Assesses stress coping skills using a 25-item self-report questionnaire that use a 5-point Likert scale from 0 to 4 (0 = strongly disagree, 4 = strongly agree). Scores range from 0 to 100, with higher scores reflecting greater resilience. Score from pre-intervention to post-intervention and 3 months follow-ups.

SECONDARY OUTCOMES:
The Ryff Scales of Psychological Well-Being - 29 items (PWBS-29; Ryff, 1989) | Up to 3 months
  Is an instrument for measuring the faces of psychological well-being, including the 6 dimensions of the Ryff model (autonomy, self-acceptance, mastery of the environment, personal growth, positive relationships with others and purpose in life). Response scores range from 1 to 6 (1 = strongly disagree, 6 = strongly agree). Score from pre-intervention to post-intervention and 3 months follow-ups.
The Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) | Up to 3 months
  Is a questionnaire to examine and diagnose patients with depressive disorders, consisting of 9 items measured on a scale of 0 to 3 (0 = not at all, 3 = almost every day). Total scores range from 0 to 27. The severity cut-off points for depression are 5, 10, 15 and 20 and represent respectively the thresholds for mild, moderate, moderately severe and severe depression. Score from pre-intervention to post-intervention and 3 months follow-ups.
Responses to Positive Affect questionnaire (RPA; Feldman et al., 2008) | Up to 3 months
  is a questionnaire that assesses the responses to positive affective states and consists of 17 items. Items are rated on a 4-point scale, ranging from 1 (almost never) to 4 (almost always). The original measure consists of three factor-analytically derived subscales: Dampening, Self-focused positive rumination, and Emotion-focused positive rumination.
Positive and Negative Effects Program (PANAS) (Watson et al., 1988) | Up to 3 months
  PANAS evaluates two independent dimensions: positive affect (PANAS+) and negative affect (PANAS-). It consists of 20 items divided into 10 range items for each dimension is from 10 to 50. Score from pre-intervention to post-intervention and 3 months follow-ups.
The Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) | Up to 3 months
  Is used to detect the presence of the symptoms of Generalized Anxiety Disorder (GAD) according to DSM-IV. It is a one-dimensional self-administered scale and although it does not provide a definitive diagnosis of GAD, it is an efficient, fast to apply, reliable and valid instrument for detecting symptoms of an anxiety disorder. The scoring scale is 0 to 3 (0 = nothing, 3 = almost every day), adding up to 0 to 21 points. They are four severity cut-off points (minimum = 0 to 4, mild = 5 to 9, moderate = 10 to 14, serious = 14 to 20) and represent the minimum to severe general anxiety thresholds. Score from pre-intervention to post-intervention and 3 months follow-ups.
The Perceived Stress Scale - 4 items (PSS-4; Cohen et al., 1983) | Up to 3 months
  Assess the extent to which recent life situations are considered stressful (Cohen et al., 1983) using a 4-item self-report questionnaire. It is a Likert scale from 1 to 5 (1 = never, 5 = very often). PSS-4 is a short version that has been used for telephone interviews or study conditions requiring short versions. Score from pre-intervention to post-intervention and 3 months follow-ups.
Self-compassion Scale - Short Form (SCS-SF; Raes et al., 2011) | Up to 3 months
  is designed to assess general self-compassion (total score) and 3 facets of this construct: common humanity (SCSCH), mindfulness (SCS-M), and self-kindness (SCS-SK) (Raes et al., 2011). This version is shorter than the original version of 26-item SCS (Neff, 2003). It contains 6 subscales representing positive and negative aspects of each facet (Raes et al., 2011). A 5-point Likert-type scale is used, ranging from 1 to 5 (1 = almost never, 5 = almost always). Score from pre-intervention to post-intervention and 3 months follow-ups.
10-Item Big Five Inventory (BFI-10; Rammstedt and John, 2007) | Up to 4 weeks
  was developed to provide a personality inventory for research environments with extreme time constraints. This questionnaire is an abridged version of the 44-item BFI. This is a 5-step scale from 1 to 5 (1 = strongly disagree, 5 = strongly agree). Score pre-intervention
The Credibility and Expectancy Questionnaire (CEQ; Devilly and Borkovec, 2000) | Up to 4 weeks
  evaluates factors of patient expectations and credibility about the treatment. This self-report consists of 6 items with answer choices rated on a 10-point scale and on a scale of 1-100%. Score pre-intervention
Client Satisfaction Questionnaire (CSQ; Attkisson and Greenfield, 1996; Larsen et al., 1979) | Up to 8 weeks
  The Client Satisfaction Questionnaire (CSQ) assesses the level of client satisfaction with health services. There are several versions of the CSQ, the longest version contains 31 items and the shortest has 8 items. The questionnaire is based on 8 questions that must be answered at the end of their stay in the service on the basis of an analogovisual scale. Each question is evaluated between 1 and 4 points and satisfaction is directly related to the number of points, so that the sum of place to a semi-quantitative variable that takes values between 8 and 32 points. The response scale is:
  csq_q1: 4=Excellent; 3=Good; 2= Regular; 1= Bad csq_q2: 1= No, definitely; 2= In very few cases; 3= Yes in general; 4=Yes definitely csq_q3: 4=Almost all; 3=Most; 2=Only a few; 1=None csq_q4: 1=No definitely; 2=No, I don't think so; 3= Yes, I think so; 4= Yes, definitely csq_q5: 1=Nothing satisfied; 2= Indifferent or moderately unsatisfied; 3=Moderately satisfied; 4=Very satisfied csq_q6: 4=If
Working Alliance Inventory for Technology Based Interventions (WAI-TECH; Kiluk et al., 2014) | Up to 8 weeks
  is a questionnaire that evaluates the therapeutic alliance between the technological tool and the patient. It covers two dimensions of the working alliance: (1) therapeutic objectives and (2) tasks. It consists of 8 items on a 5-point Likert scale from 1 to 5 (1 = never, 5 = always). Score from post-treatment
Overall Anxiety Severity and Impairment Scale (OASIS; Norman et al. 2006) | Up to 8 weeks
  It is a 5-item questionnaire, with a score of 0 to 4, that evaluates the frequency and severity of anxiety symptoms. The instrument also provides measures related to anxiety symptoms such as avoidance, work, academy, social and daily life disabilities. According to a psychometric analysis it has good internal consistency (α =.80), test-test reliability (k =.82) and convergent validity. Score from pre-intervention to post-intervention
Overall Depression Severity and Impairment Scale (ODSIS; Bentley, et. Al 2014). | Up to 8 weeks
  It is a self-report measure with five items that assess experiences related to depression, measuring its frequency and severity, as well as the level of avoidance behaviors, interference between work, school and home, and associated social. The internal consistency of the scale has proven to be excellent, with a Cronbach alpha between 0.91 and 0.94 and good convergent and discriminant validity. Score from pre-intervention to post-intervention
Openness to the future Scale (OF)(Botella et a.l, 2018 ) | Up to 3 months
  It is a scale consisting of 10 items of scores ranging from 1 to 5 on a likert scale and assesses expectations and positive affectivity towards the future, which includes five domains: (1) Illusion of control (2) Acceptance (3) Commitment to life and planning (4) Positive orientation towards the future (5) Self-efficacy towards the future.

OTHER OUTCOMES:
Socio-demographic data | Up to 4 weeks
  Measurements of sociodemographic variables are included: sex, household size and income, age, marital status, employment status, total population of the place of residence, nationality, level of education and living situation. In addition, health-related variables will be measured: presence of psychological disorders (past and present) and whether treatment is currently being carried out. Score from pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, PhD, Study Director — University Jaume I, Castellon, Spain; Araceli Palma Gómez, Phd Student, Principal Investigator — University Jaume I, Castellon, Spain; Rocio Herrero, PhD, Principal Investigator — University Jaume I, Castellon, Spain
Locations (5):
- Argentina (2):
  - Universidad de Mar del Plata, Mar del Plata, Buenos Aires
  - Universidad de Buenos Aires, Buenos Aires
- Universidad Autónoma del Estado de Hidalgo, Pachuca, Hidalgo, Mexico
- Spain (2):
  - Univesity Jaume I, Castellon, Castellon
  - Universitat de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banos RM, Etchemendy E, Mira A, Riva G, Gaggioli A, Botella C. Online Positive Interventions to Promote Well-being and Resilience in the Adolescent Population: A Narrative Review. Front Psychiatry. 2017 Jan 30;8:10. doi: 10.3389/fpsyt.2017.00010. eCollection 2017. PMID 28194117
- [Background] Cuijpers P, Cristea IA, Ebert DD, Koot HM, Auerbach RP, Bruffaerts R, Kessler RC. PSYCHOLOGICAL TREATMENT OF DEPRESSION IN COLLEGE STUDENTS: A METAANALYSIS. Depress Anxiety. 2016 May;33(5):400-14. doi: 10.1002/da.22461. Epub 2015 Dec 18. PMID 26682536
- [Background] Ryff CD. Psychological well-being revisited: advances in the science and practice of eudaimonia. Psychother Psychosom. 2014;83(1):10-28. doi: 10.1159/000353263. Epub 2013 Nov 19. PMID 24281296
- [Background] Salamanca-Sanabria A, Richards D, Timulak L, Castro-Camacho L, Mojica-Perilla M, Parra-Villa Y. Assessing the efficacy of a culturally adapted cognitive behavioural internet-delivered treatment for depression: protocol for a randomised controlled trial. BMC Psychiatry. 2018 Feb 27;18(1):53. doi: 10.1186/s12888-018-1634-x. PMID 29482586
- [Background] Leppin AL, Bora PR, Tilburt JC, Gionfriddo MR, Zeballos-Palacios C, Dulohery MM, Sood A, Erwin PJ, Brito JP, Boehmer KR, Montori VM. The efficacy of resiliency training programs: a systematic review and meta-analysis of randomized trials. PLoS One. 2014 Oct 27;9(10):e111420. doi: 10.1371/journal.pone.0111420. eCollection 2014. PMID 25347713
- [Background] Dray J, Bowman J, Campbell E, Freund M, Hodder R, Wolfenden L, Richards J, Leane C, Green S, Lecathelinais C, Oldmeadow C, Attia J, Gillham K, Wiggers J. Effectiveness of a pragmatic school-based universal intervention targeting student resilience protective factors in reducing mental health problems in adolescents. J Adolesc. 2017 Jun;57:74-89. doi: 10.1016/j.adolescence.2017.03.009. Epub 2017 Apr 3. PMID 28384523
- [Background] Ebert DD, Zarski AC, Christensen H, Stikkelbroek Y, Cuijpers P, Berking M, Riper H. Internet and computer-based cognitive behavioral therapy for anxiety and depression in youth: a meta-analysis of randomized controlled outcome trials. PLoS One. 2015 Mar 18;10(3):e0119895. doi: 10.1371/journal.pone.0119895. eCollection 2015. PMID 25786025
- [Background] Ibrahim AK, Kelly SJ, Adams CE, Glazebrook C. A systematic review of studies of depression prevalence in university students. J Psychiatr Res. 2013 Mar;47(3):391-400. doi: 10.1016/j.jpsychires.2012.11.015. Epub 2012 Dec 20. PMID 23260171
- [Background] Day V, McGrath PJ, Wojtowicz M. Internet-based guided self-help for university students with anxiety, depression and stress: a randomized controlled clinical trial. Behav Res Ther. 2013 Jul;51(7):344-51. doi: 10.1016/j.brat.2013.03.003. Epub 2013 Mar 28. PMID 23639300
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879
- [Derived] Palma-Gomez A, Herrero R, Banos R, Garcia-Palacios A, Castaneiras C, Fernandez GL, Llull DM, Torres LC, Barranco LA, Cardenas-Gomez L, Botella C. Efficacy of a self-applied online program to promote resilience and coping skills in university students in four Spanish-speaking countries: study protocol for a randomized controlled trial. BMC Psychiatry. 2020 Apr 5;20(1):148. doi: 10.1186/s12888-020-02536-w. PMID 32248795
- See also: Psychology and Technology is a platform that contains treatment programs for different mental and physical health problems, which can be applied according to the specific needs of each person, step by step, and adapting to the pace of the user, from home — https://psicologiaytecnologia.labpsitec.es/